CLINICAL TRIAL: NCT00002277
Title: Fluconazole Versus Amphotericin B: A Prospective, Randomized, Multicenter Study for Therapy of Fungal Infection
Brief Title: A Comparison of Fluconazole and Amphotericin B in the Treatment of Fungal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012N; 056-173
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-12

CONDITIONS: Mycoses; HIV Infections
Keywords: Mycoses; Neoplasms; Neutropenia; Fluconazole; Amphotericin B
MeSH Terms: conditions — Mycoses; HIV Infections; Neoplasms; Neutropenia | interventions — Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety, tolerance and efficacy of fluconazole and amphotericin B as treatment for biopsy proven fungal infections in major organs, disseminated infection, suspected fungal infection and fungemia in adult neutropenic and non-neutropenic patients without AIDS, AIDS related complex (ARC), or extensive burns. HIV seropositive patients are allowed only if they also have a malignancy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunostimulants under studies carried out under an IRB approved protocol.
* Treatments of intercurrent non-fungal infection.
* Allowed but requires monitoring during fluconazole therapy:
* Barbiturates.
* Phenytoin.
* Oral hypoglycemics.
* Coumarin-type anticoagulants.

Patients must have the following:

* Diagnosis or presumption of fungal infection under defined conditions.
* Written informed consent either from the patient or the patient's legal guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Burns > 30 percent of the body.
* Diagnosis of AIDS or AIDS related complex (ARC).
* HIV positive unless they have a malignancy.
* History of allergy to or intolerance of imidazoles or azoles.
* Moderate to severe liver disease as defined by specific lab values.
* Unlikely to survive more than 24 hours.
* Evidence of previous amphotericin B sensitivity.

Concurrent Medication:

Excluded:

* Concomitant antifungal agents other than the study drugs.
* Immunostimulants, except for studies carried out under an IRB approved protocol.

Concurrent Treatment:

Excluded:

* Lymphocyte replacements.

Patients with the following are excluded:

* Defined disease conditions listed in Exclusion Co-Existing Conditions.
* Unlikely to survive more than 24 hours.
* Previous participation in this study; reentry for the same infection is not allowed.
* Known to be unable to take amphotericin B due to acute toxicities.

Prior Medication:

Excluded:

* Previous fluconazole therapy for this infection.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dr Layne Gentry, Houston, Texas
  - Dr Temple Williams, Houston, Texas
  - M D Anderson Cancer Ctr, Houston, Texas